CLINICAL TRIAL: NCT04935840
Title: Clinical Study to Evaluate the Effect of a Food Supplement With Probiotics on the Metabolic Profile of Pregnant Women
Brief Title: Evaluation of the Effect of FertyBiotic Pregnancy in the Metabolic Profile in Pregnant Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fertypharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020_FBE_04
Record Dates: First submitted 2021-06-07; First posted 2021-06-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FertyBiotic Pregnancy (Experimental): Participants received FertyBiotic Pregnancy one capsule a day
  Interventions: Dietary Supplement: FertyBiotic Pregnancy; Other: Control

INTERVENTIONS:
Dietary Supplement: FertyBiotic Pregnancy — DHA, folic acid, Iodine, iron, Lactobacillus rhamnosus, Lactobacillus reuterii, magnesium, zinc, vitamin D3, Vitamin C, Vitamin E, Group B vitamins and Biotin
Other: Control — 400 mcg of folic acid

SUMMARY:
The aim of this study is determine the effect of a food supplement with probiotics on metabolic profile and weight gain in pregnant women.

DETAILED DESCRIPTION:
After being informed about the study, all patients meeting the inclusion/exclusion criteria and giving written informed consent all patients will be treated with the food supplement that contain vitamins, minerals and probiotics. All volunteers will receive one capsule per day of the food supplement throughout the study. The duration of the supplementation will be from their inclusion in the study (≤ 14 weeks of gestation) until the 30th-32nd week of pregnancy, the time of the end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age: > 18 years old
* BMI > 25
* Women who have signed the informed consent to participate in the study.
* No intention to change their routine physical activity or usual dietary intakes throughout the study

Exclusion Criteria:

* > 14 weeks' gestation
* Taking food supplements or probiotics
* History or current pathology that influence in the study
* With major fetal abnormalities
* Had used continuous antibiotic therapy for at least 3 months

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 84 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-03-23 (Estimated)

PRIMARY OUTCOMES:
Glucose homeostasis | 30-32 weeks gestation
  Glucose homeostasis status will be evaluated by measuring fasting glucose

SECONDARY OUTCOMES:
Insulin levels | 30-32 weeks gestation
  Insulin levels status will be evaluated by measuring fasting insulin
Insulin resistance | 30-32 weeks gestation
  Insulin resistance will be evaluated by measuring HOMA IR and QUICKI index (fasting glucose and fasting insulin combination)
Weight gain | 30-32 weeks gestation
  Weight will be evaluated weighting the subjects
Lipid concentration | 30-32 weeks gestation
  Lipid concentration will be evaluated by measuring fasting total colesterol, LDL, HDL and triglyceride

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Vithas Medimar, Alicante, Alicante
  - Centro Ginecologico Dra. García-Pérez Llantada, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No